CLINICAL TRIAL: NCT03184467
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Design, Prospective, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Donepezil and Combined With GV1001 in Alzheimer Patients
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of GV1001 in Alzheimer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GemVax & Kael (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KG 6/2016
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease
Keywords: GV1001; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Normal saline 0.9%
  Interventions: Drug: Normal Saline 0.9%
- Study group 1 (Experimental): GV1001 0.56 mg
  Interventions: Drug: GV1001 0.56 mg
- Study group 2 (Experimental): GV1001 1.12 mg
  Interventions: Drug: GV1001 1.12 mg

INTERVENTIONS:
Drug: Normal Saline 0.9% — Normal saline 0.9% is subcutaneously administered once weekly schedule for 4 weeks (4 times) followed by every two weeks until week 24 (10 times). A total number of administration is 14 times.
  Other Names: NS 0.9%
  Arms: Control group
Drug: GV1001 0.56 mg — GV1001 0.56 mg is subcutaneously administered once weekly schedule for 4 weeks (4 times) followed by every two weeks until week 24 (10 times). A total number of administration is 14 times.
  Other Names: Tertomotide
  Arms: Study group 1
Drug: GV1001 1.12 mg — GV1001 1.12 mg is subcutaneously administered once weekly schedule for 4 weeks (4 times) followed by every two weeks until week 24 (10 times). A total number of administration is 14 times.
  Other Names: Tertomotide
  Arms: Study group 2

SUMMARY:
This clinical study is designed as a multi-center, randomized, double-blind, placebo-controlled, parallel design, prospective, phase II clinical trial.

An eligible subject who meets inclusion and exclusion criteria is randomly assigned to three groups: study group 1 (GV1001 0.56 mg), study group 2 (GV1001 1.12 mg) or placebo group. A randomized subject is administered either GV1001 or placebo in a total of 14 times and will be evaluated for the efficacy and safety at week of 24.

DETAILED DESCRIPTION:
GV1001 0.56 mg, 1.12 mg or placebo is subcutaneously administered once weekly schedule for 4 weeks (4 times) followed by every two weeks until week 24 (10 times). A total number of administration is 14 times.

1. Control group (placebo): 30 subjects
2. Study group 1 (GV1001 0.56 mg): 30 subjects
3. Study group 2 (GV1001 1.12 mg): 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 55 to 85 years of age
2. A patient who satisfies diagnostic criteria for dementia in DSM-IV
3. Probable Alzheimer's disease in NINCDS-ADRDA
4. K-MMSE ≤ 19 at screening and randomization visit
5. GDS 5~6 stage
6. MRI or CT scan within 12 months prior to screening visit that proves Alzheimer's disease without any other disease that may cause dementia
7. A patient taking stable doses of donepezil for more than 3 months before screening visit
8. A patient who are able to visit a hospital (including inpatient and outpatient based) and receive cognitive and other tests
9. A patient with a caregiver who can accompany all visits and supervise the subject's compliance with the procedures and study drug prescribed in the protocol, and provide detailed information about the patient
10. Written informed consent by a patient or legal representative

Exclusion Criteria:

1. Any other cause of dementia shown by CT / MRI findings and neurological examination within 12 months of screening visit

   * Possible, probable or definite vascular dementia according to the NINDS-AIREN
   * Other central nervous system diseases that may cause cognitive impairment (cerebrovascular disease including cerebrovascular dementia, Parkinsonism, Huntington's disease, subdural hematoma, normal pressure hydrocephalus, brain tumor, Creutzfeldt-Jakob disease, etc.)
   * Neurological deficits such as delusions, delirium, epilepsy
2. Vitamin B12, folic acid, syphilis serology, and thyroid stimulating hormone (TSH) results are thought to contribute to the severity of dementia or cause dementia
3. A patient who are considered ineligible for this study by investigator due to concurrent or history of significant psychiatric conditions (eg. schizophrenia or bipolar affective disorder)
4. A patient with a history of known or suspected seizures including febrile seizures, a history of significant head trauma with loss of consciousness or recent unconsciousness that is not explained
5. A patient with acute or unstable cardiovascular disease, active peptic ulcer, uncontrolled hypertension, uncontrolled diabetes or insulin dependent patients or any medical condition that may interfere with the completion of clinical trials
6. Hypersensitivity to investigational medicinal products
7. History of alcohol, substance abuse or dependence (except nicotine dependence) within the last 2 years
8. Concurrent malignancies or invasive cancers diagnosed within the past 5 years except for non-metastatic basal cell carcinoma or squamous cell carcinoma of skin, in situ carcinoma of the uterine cervix or non-metastatic prostate cancer
9. Renal impairment (creatinine clearance (CLcr) <30 mL / min)
10. Severe liver dysfunction (ALT or AST> 2 times the upper limit of normal)
11. A patient taking other drugs other than donepezil to treat Alzheimer's disease or other cognitive impairment
12. A patient taking other drugs other than anticholinergic drugs, cholinergic drugs (local usages are allowable, such as pilocarpine eye drops), antidepressants (tricyclic antidepressant, MAO inhibitor) antipsychotics, donepezil to treat Alzheimer's disease
13. Women at childbearing age who do not consent using medicinally acceptable contraception (such as surgical sterilization, intrauterine contraceptive device, condom or diaphragm, an injectable or inserted contraceptive) during the study
14. Pregnancy or breast feeding
15. A patient who participated in other clinical trials within 4 weeks prior to this study
16. 35 kg weight or below
17. A patient who had experienced this study drug
18. A patient who had participated in a clinical trial for Alzheimer dementia vaccine within last 6 months
19. Any other patients who are considered to be ineligible for this study by an investigator

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
SIB (Severe Impairment Battery) | week 24
  Change in SIB compared to the baseline and week 24

SECONDARY OUTCOMES:
K-MMSE (Korean-Mini-Mental State Examination) | week 24
  Change in K-MMSE compared to the baseline and week 24
CDR-SOB (Clinical Dementia Rating-Sum of Box) | week 24
  Change in CDR-SOB compared to the baseline and week 24
NPI (Neuropsychiatric Inventory) | week 24
  Change in NPI compared to the baseline and week 24
GDS (Global Deterioration Scale) | week 24
  Change in GDS compared to the baseline and week 24
ADCS-ADL-severe (Alzheimer's Disease Cooperative Study-Activities of Daily Living scale-severe) | week 24
  Change in ADCS-ADL-severe compared to the baseline and week 24
CIBIC-plus (Clinician Interview-Based Impression of Change-Plus) | week 24
  Change in CIBIC-plus compared to the baseline and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Gon Song, MD., PhD., Study Director — GemVax & Kael
Locations (1):
- Hanyang University Guri Hospital, Guri-si, Gyunggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kwon HS, Koh SH, Choi SH, Jeong JH, Na HR, Lee CN, Yang Y, Lee AY, Lee JH, Park KW, Han HJ, Kim BC, Park J, Lee JY, Lee KY, Kim S. Effects of GV1001 on Language Dysfunction in Patients With Moderate-to-Severe Alzheimer's Disease: Post Hoc Analysis of Severe Impairment Battery Subscales. Dement Neurocogn Disord. 2023 Jul;22(3):100-108. doi: 10.12779/dnd.2023.22.3.100. Epub 2023 Jul 11. PMID 37545861
- [Derived] Koh SH, Kwon HS, Choi SH, Jeong JH, Na HR, Lee CN, Yang Y, Lee AY, Lee JH, Park KW, Han HJ, Kim BC, Park JS, Lee JY, Kim S, Lee KY. Efficacy and safety of GV1001 in patients with moderate-to-severe Alzheimer's disease already receiving donepezil: a phase 2 randomized, double-blind, placebo-controlled, multicenter clinical trial. Alzheimers Res Ther. 2021 Mar 26;13(1):66. doi: 10.1186/s13195-021-00803-w. PMID 33771205